CLINICAL TRIAL: NCT01195519
Title: The Study Will Investigate the Quality of Life in PD or HD Patients
Brief Title: The Assessment of Quality of Life in Patients With Peritoneal Dialysis and Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Tso-Hsiao Chen, Nephrology Dean
Other Study IDs: 99039
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Peritoneal Dialysis; Hemodialysis
Keywords: peritoneal dialysis; hemodialysis patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- peritoneal dialysis and hemodialysis patients: peritoneal dialysis and hemodialysis patients

SUMMARY:
Currently, lots of researches aimed at quality of life of patients with peritoneal dialysis and hemodialysis related issues. There is no study related to establish the predictive model of quality of life. This study will investigate the predictive model of quality of life in terms of peritoneal dialysis (PD) or hemodialysis (HD) patients. These results will offer the further evidence to the government to develop the effective interventions for dialysis patients. The optimal goal is to promote the quality care.

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old PD or HD patients
* conscious clear and no psychosis
* literate and can communicate
* willing to participate and sign informed consent

Exclusion Criteria:

* Not volunteer
* subject felt weak or uncomfortable and patients decision to withdraw from the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: peritoneal dialysis and hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2010-09; Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tso-Hsiao Chen, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, No.111, Section 3, Hsing-Long Rd, Taipei, Taiwan

REFERENCES:
- See also: Click here for more information about this study — http://www.wanfang.gov.tw/